CLINICAL TRIAL: NCT02177123
Title: Post Market Study to Evaluate Safety and Effectiveness of the InnFocus Microshunt™ (MIDI Arrow) in Patients With Primary Open Angle Glaucoma
Brief Title: Post Market Study of the InnFocus MicroShunt
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: InnFocus Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: INN-007
Record Dates: First submitted 2014-06-26; First posted 2014-06-27 (Estimated); Results first posted 2021-05-28 (Actual); Last update posted 2021-06-24 (Actual); Status verified 2021-06

CONDITIONS: Primary Open Angle Glaucoma
Keywords: glaucoma shunt; glaucoma drainage device
MeSH Terms: conditions — Glaucoma, Open-Angle

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- InnFocus MicroShunt Surgery (Experimental): InnFocus MicroShunt implantation in the anterior chamber of the eye on patients with primary open angle glaucoma after am antiproliferative treatment of mitomycin C (MMC)
  Interventions: Device: InnFocus MicroShunt implantation

INTERVENTIONS:
Device: InnFocus MicroShunt implantation — Implantation will include the use of Mitomycin C applied with sponges.
  Other Names: InnFocus MicroShunt; MIDI Arrow

SUMMARY:
Prospective, multicentric, single arm post market study to gather safety and effectiveness data on the CE Marked InnFocus MicroShunt (MIDI Arrow) device in primary open angle glaucoma patients

DETAILED DESCRIPTION:
The purpose of this study is to collect additional safety and effectiveness data on the InnFocus MicroShunt (MIDI Arrow) in subjects suffering from primary open angle glaucoma who are inadequately controlled on maximum tolerated medical therapy with intraocular pressure ≥ 18 mm Hg and ≤ 35 mm Hg and/or where glaucoma progression warrants surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Subject has mild to moderate primary open glaucoma where the intraocular pressure is not adequately controlled on maximum tolerated medical therapy and has intraocular pressure greater than or equal to 18mmHg and less than or equal to 35mmHg while on glaucoma medications and/or where glaucoma progression warrants surgery.
2. Primary open angle glaucoma diagnosis based on glaucomatous optic nerve damage as evidenced by any of the following optic disc or retinal nerve fiber layer structural abnormalities documented on slit lamp stereo biomicroscopy or in stereo disc photos:

   1. Diffuse thinning, focal narrowing, or notching of the optic disc rim, especially at the inferior or superior poles.
   2. Localized abnormalities of the peripapillary retinal nerve fiber layer, especially at the inferior or superior poles.
   3. Optic disc neural rim asymmetry of the two eyes consistent with loss of neural tissue.
   4. Disc rim or peripapillary retinal nerve fiber layer hemorrhages.

4) Subject willing to comply with study requirements. 5) Subject who has signed an approved informed consent form

Exclusion Criteria:

1. Active iris neovascularization, active proliferative retinopathy or other ophthalmic disease that could confound study results.
2. Iridocorneal endothelial syndrome.
3. Epithelial or fibrous downgrowth.
4. Secondary glaucoma such as post-trauma, pseudo-exfoliative, etc.
5. Chronic ocular inflammatory disease.
6. Prior argon laser, selective laser, or micropulse trabeculoplasty within 90 days of enrollment.
7. Inability to obtain accurate IOP measurement throughout the study. For example: a history of corneal surgery, corneal opacities or disease/pathology (Active corneal infection or Fuchs dystrophy are examples.).
8. Severe anterior or posterior blepharitis.
9. Previous incisional ophthalmic surgery, excluding uncomplicated clear corneal phacoemulsification (cataract) surgery at least 6 months prior to enrollment.
10. Prior laser peripheral iridotomy.
11. Fellow eye with poorer than 20/200 best-corrected visual acuity (BCVA)
12. Angle closure glaucoma or narrow anatomical chamber angle as identified by gonioscopy and classified as Shaffer Grade 0 or 1.
13. Previous cyclodestructive procedure.
14. Use of oral hypotensive glaucoma medications for treatment of the fellow eye.
15. Severe anterior or posterior blepharitis.
16. Unwilling to discontinue contact lens use after surgery.
17. Previous incisional ophthalmic surgery, excluding uncomplicated clear corneal phacoemulsification (cataract) surgery at least 6 months prior to enrollment.
18. Presence of an anterior chamber IOL (AC-IOL).
19. Prior laser peripheral iridotomy.
20. Need for glaucoma surgery combined with other ocular procedures or anticipated need for additional ocular surgery during the investigational period.
21. Fellow eye with poorer than 20/200 best-corrected visual acuity (BCVA)
22. Known allergy or other contraindication to Mitomycin C (MMC) drug.
23. Angle closure glaucoma or narrow anatomical chamber angle as identified by gonioscopy and classified as Shaffer Grade 0 or 1.
24. Any condition that prevents the investigational device implantation or trabeculectomy in the superior region of the study eye (e.g., peripheral anterior synechiae, scleral staphyloma or conjunctival scarring).
25. Diagnosed degenerative visual disorders not associated with existing glaucoma condition (e.g., advanced dry or wet macular degeneration or other retinal disorders, central retinal artery or vein occlusion) or choroidopathy (e.g., choroidal detachment, effusion, choroiditis, or neovascularization).
26. Central corneal thickness that is less than 450 microns or greater than 620 microns.
27. Previous cyclodestructive procedure.
28. Prior retinal laser procedure conducted for any purpose other than treatment of retinal tear or hole.
29. Conditions associated with elevated episcleral venous pressure such as active thyroid orbitopathy, cavernous sinus fistula, Sturge-Weber syndrome, orbital tumors, orbital congestive disease.
30. Clinically significant sequelae from trauma (e.g., chemical burns, blunt trauma, etc.)
31. Ocular pathology or medical condition for which, in the investigator's judgment, the following factors would either place the subject at increased risk of complications or contraindicate device implantation or interfere with compliance to elements of the study protocol (e.g., ophthalmic examinations, follow-up visits),

    1. inability to reliably complete visual field testing over the course of the study,
    2. uncontrolled systemic disease (e.g. diabetes, hypertension) that could compromise their participation in the study.
    3. Disorders that pose a fall risk, as well as compromise ability to take a visual field exam and take glaucoma medications (e.g., Parkinson's disease),
    4. inability to discontinue use of blood thinners within the surgeon's standard preoperative or postoperative instructions.
    5. immunodeficiency concerns.
    6. known corticosteroid responders whose pressure increases would not allow them to withstand the postop corticosteroid regimen.
32. Intraocular silicone oil.
33. Ocular steroid use in the planned study eye or systemic steroid use anytime within three months of the procedure. (This would not include the use of inhaled or dermatologic steroids.)
34. Chemotherapy within six months of the screening visit.
35. Use of oral hypotensive glaucoma medications for treatment of the fellow eye.
36. A requirement of general anesthesia for the procedure.
37. Bacterial conjunctivitis
38. Bacterial corneal ulcers
39. Endophthalmitis
40. Orbital cellulitis
41. Bacteremia or septicemia
42. Active scleritis
43. Uveitis
44. Severe dry eye syndrome
45. Severe myopia
46. Pseudo-exfoliative glaucoma

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2014-04-04 (Actual); Primary Completion 2017-11-27 (Actual); Study Completion 2017-11-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Guy Van de Weyer, Optometrist, Study Director — InnFocus Inc.
Locations (6):
- France (3):
  - Clinique Ophtalmologique Universitaire de Grenoble, Hôpital A. Michallon - CHU de Grenoble, Grenoble
  - Groupe hospitalier Paris Saint-Joseph, Service d'Ophtalmologie, Paris
  - Pole Ophtalmologique de la Clinique Mutualiste, Pessac
- University Eye Clinic Maastricht, Maastricht, Netherlands
- Clinicovision - Hospital Clinico San Carlos, Madrid, Spain
- Hôpitaux Universitaires de Genève, Policlinique d'Ophtalmologie, Geneva, Switzerland

REFERENCES:
- [Derived] Garcia-Feijoo J, Batlle JF, Aptel F, Lachkar Y, Riss I, Sadruddin O, Nguyen T, Beckers HJM. Pooled Analysis of Three MicroShunt Studies in Primary Open-Angle Glaucoma Evaluating Different Concentrations of Applied Mitomycin C. Ophthalmol Ther. 2025 Jul;14(7):1533-1549. doi: 10.1007/s40123-025-01149-4. Epub 2025 May 23. PMID 40408035
- [Derived] Beckers HJM, Aptel F, Webers CAB, Bluwol E, Martinez-de-la-Casa JM, Garcia-Feijoo J, Lachkar Y, Mendez-Hernandez CD, Riss I, Shao H, Pinchuk L, Angeles R, Sadruddin O, Shaarawy TM. Safety and Effectiveness of the PRESERFLO(R) MicroShunt in Primary Open-Angle Glaucoma: Results from a 2-Year Multicenter Study. Ophthalmol Glaucoma. 2022 Mar-Apr;5(2):195-209. doi: 10.1016/j.ogla.2021.07.008. Epub 2021 Jul 28. PMID 34329772

RESULTS

PARTICIPANT FLOW:
Groups:
- Subjects Suffering From Primary Open Angle Glaucoma: Subjects suffering from primary open angle glaucoma who are inadequately controlled on maximum tolerated medical therapy with intraocular pressure ≥ 18 mm Hg and ≤ 35 mm Hg and/or.where glaucoma progression warrants surgery
Period: Overall Study
Arm/Group | Subjects Suffering From Primary Open Angle Glaucoma
Started | 107
Completed | 83
Not Completed | 24
Not completed — Lost to Follow-up | 6
Not completed — Withdrawal by Subject | 4
Not completed — Adverse Event | 4
Not completed — Physician Decision | 3
Not completed — Excluded by Sponsor - other reason | 2
Not completed — Excluded for medical reasons | 2
Not completed — Death | 1
Not completed — Other | 1
Not completed — Excl. #31 Ocular pathology or medical condition which would place subject at increased risk | 1

BASELINE CHARACTERISTICS:
Population: The Intent-to-Treat (ITT) population included all patients who have signed the informed consent and received the assigned therapy under evaluation (InnFocus MicroShunt).
Arm/Group | Subjects Suffering From Primary Open Angle Glaucoma
Number analyzed (Participants) | 101
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.7 (12.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 53
  Male | 48
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  France | 65
  Switzerland | 8
  Netherlands | 12
  Spain | 16

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Study Success
Description: Rate of success with respect to IOP at Months 6, 9, 12 and 24 on ITT population
Time Frame: Month 6, 9, 12, and 24
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Groups:
- Success With Respect for IOP: The rates of success reflected sustained control of IOP
Arm/Group | Success With Respect for IOP
Number analyzed (Participants) | 101
Participants
  Month 6 | 62
  Month 9 | 59
  Month 12 | 58
  Month 24 | 60

2. Secondary Outcome: IOP Change
Description: IOP relative to the pre-operative value was assessed at each post-operative visit (Day 1, Day 7, Week 4, Month 3, Month 6, Month 9, Month 12, and Month 24).
Time Frame: Day 1, Day 7, Week 4, Month 3, Month 6, Month 9, Month 12, and Month 24
Population: The Intent-to-Treat (ITT) population included all patients who have signed the informed consent and received the assigned therapy under evaluation (InnFocus MicroShunt).
  IOP data collected after glaucoma re-operation was censored for this analysis.
Measure: Mean (Standard Deviation); unit: mmHg
Groups:
- IOP Changes From Baseline: IOP Changes from Baseline thur all timepoints
Arm/Group | IOP Changes From Baseline
Number analyzed (Participants) | 101
mmHg
  Baseline | 21.5 (4.2)
  Day 1: number analyzed (Participants) | 97
  Day 1 | 9.5 (2.9)
  Day 7: number analyzed (Participants) | 97
  Day 7 | 9.8 (3.5)
  Week 4: number analyzed (Participants) | 98
  Week 4 | 12.8 (6.0)
  Month 3: number analyzed (Participants) | 93
  Month 3 | 14 (5.2)
  Month 6: number analyzed (Participants) | 87
  Month 6 | 15 (4.7)
  Month 9: number analyzed (Participants) | 78
  Month 9 | 15.3 (6.6)
  Month 12: number analyzed (Participants) | 78
  Month 12 | 15 (4)
  Month 24: number analyzed (Participants) | 71
  Month 24 | 14 (3)

3. Other Pre Specified Outcome: Number of Participants Requiring Supplemental Medical Therapy at M12 and M24
Description: Throughout the study, the number of glaucoma supplemental medications (derived as the number of medication classes) required after the IMS procedure.
Time Frame: 12 and 24 Months
Population: Patients Taking Glaucoma Supplemental Treatment (Study Eye) ITT
Measure: Count of Participants; unit: Participants
Groups:
- Need for Glaucoma Supplemental Treatment at M12; Need for Glaucoma Supplemental Treatment at M24: Patients Taking Glaucoma Supplemental Treatment (Study Eye)
Arm/Group | Need for Glaucoma Supplemental Treatment at M12 | Need for Glaucoma Supplemental Treatment at M24
Number analyzed (Participants) | 78 | 71
Participants | 25 | 25

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were reported for the duration of the study (approximatively 36 months). This analysis population includes all patients who have signed the informed consent / enrolled in the study.
Description: Any untoward medical occurrence, unintended disease or injury or any untoward clinical signs (including an abnormal laboratory finding) in subjects, users or other persons whether or not related to the investigational medical device.
Arm/Group | Subjects Suffering From Primary Open Angle Glaucoma
All-Cause Mortality (participants affected / at risk) | 1/107
Serious Adverse Events (participants affected / at risk) | 11/107
Other Adverse Events (participants affected / at risk) | 67/107
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Subjects Suffering From Primary Open Angle Glaucoma (N=107)
Allergic Keratitis (Eye disorders) | 1 (1)
Anterior Chamber Inflammation (Eye disorders) | 1 (1)
Cataract (Eye disorders) | 1 (1)
Ulcerative Keratitis (Eye disorders) | 1 (1)
Intraocular Pressure Increased (Investigations) | 4 (4)
Sclerectomy (Surgical and medical procedures) | 1 (1)
Trabeculectomy (Surgical and medical procedures) | 1 (1)
Implant Site Dehiscence (General disorders) | 1 (2) — and administration site conditions
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Subjects Suffering From Primary Open Angle Glaucoma (N=107)
Hypotony Of Eye (Eye disorders) | 10 (10)
Conjunctival Bleb (Eye disorders) | 8 (10)
Keratitis (Eye disorders) | 8 (8)
Lacrimation Increased (Eye disorders) | 5 (6)
Cataract (Eye disorders) | 4 (5)
Eye Pain (Eye disorders) | 4 (5)
Punctate Keratitis (Eye disorders) | 4 (4)
Visual Acuity Reduced (Eye disorders) | 5 (5)
Hyphaema (Eye disorders) | 4 (4)
Vision Blurred (Eye disorders) | 2 (2)
Eyelid Ptosis (Eye disorders) | 3 (3)
Flat Anterior Chamber Of Eye (Eye disorders) | 3 (3)
Ulcerative Keratitis (Eye disorders) | 2 (2)
Diplopia (Eye disorders) | 2 (2)
Dry Eye (Eye disorders) | 2 (2)
Eye Inflammation (Eye disorders) | 1 (1)
Eye Pruritus (Eye disorders) | 1 (2)
Allergic Keratitis (Eye disorders) | 1 (1)
Anterior Chamber Inflammation (Eye disorders) | 1 (1)
Choroidal Effusion (Eye disorders) | 1 (1)
Conjunctival Haemorrhage (Eye disorders) | 1 (1)
Conjunctival Hyperaemia (Eye disorders) | 1 (1)
Conjunctival Ulcer (Eye disorders) | 1 (1)
Corneal Oedema (Eye disorders) | 1 (1)
Iris Adhesions (Eye disorders) | 1 (1)
Posterior Capsule Opacification (Eye disorders) | 1 (1)
Intraocular Pressure Increased (Investigations) | 26 (35)
Implant Site Dehiscence (General disorders) | 6 (8)
Pain (General disorders) | 2 (2)
Complication Of Device Insertion (General disorders) | 1 (1)
Encapsulation Reaction (General disorders) | 1 (1)
Conjunctival Filtering Bleb Leak (Injury, poisoning and procedural complications) | 2 (2)
Anaesthetic Complication (Injury, poisoning and procedural complications) | 1 (1)
Suture Related Complication (Injury, poisoning and procedural complications) | 2 (2)
Post Procedural Complication (Injury, poisoning and procedural complications) | 1 (1)
Tenon's Cyst (Injury, poisoning and procedural complications) | 1 (1)
Cataract Operation (Surgical and medical procedures) | 1 (1)
Sclerectomy (Surgical and medical procedures) | 2 (2)
Trabeculectomy (Surgical and medical procedures) | 1 (1)
Conjunctivitis (Infections and infestations) | 2 (2)
Hordeolum (Infections and infestations) | 1 (1)
Device Dislocation (Product Issues) | 2 (2)
Device Occlusion (Product Issues) | 1 (1)
Needle Issue (Product Issues) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2015-03-09): https://cdn.clinicaltrials.gov/large-docs/23/NCT02177123/Prot_000.pdf
  • Statistical Analysis Plan (2018-03-05): https://cdn.clinicaltrials.gov/large-docs/23/NCT02177123/SAP_001.pdf